CLINICAL TRIAL: NCT02173600
Title: Estimation of Cardiovascular Risk After Intensive Dietary Counselling in a Primary Care Setting
Brief Title: Cardiovascular Risk Factors And Intensive Dietary Counselling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Andalusian Regional Ministry of Health (Other Government)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Dr. María Ángeles Rubín-Gómez, Dr, Andalusian Regional Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-0969-12
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: High Blood Pressure; Hypercholesterolemia; Tobacco Smoking
Keywords: Cardiovascular risk; Primary prevention; Intensive dietary counselling; Physical exercise
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Tobacco Smoking; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group-level Intensive Dietary Counselling (Experimental): Active learning through 4-6 60-minute sessions workshop, enrolling 8-12 people each time.
  Interventions: Behavioral: Group-level Intensive dietary Counselling
- Individual-level Intensive Dietary Counselling (Active Comparator): Individualised dietary counselling delivered at the health-care point
  Interventions: Behavioral: Individual-level Intensive Dietary Counselling

INTERVENTIONS:
Behavioral: Group-level Intensive dietary Counselling
  Arms: Group-level Intensive Dietary Counselling
Behavioral: Individual-level Intensive Dietary Counselling
  Arms: Individual-level Intensive Dietary Counselling

SUMMARY:
The Intensive Dietary Counselling (IDC) intervention is a prevention and health promotion activity. It is being implemented by the Andalusian Health Service to reinforce basic intervention advice on healthy diet and exercise. The IDC intervention is aimed at the prevention of diseases of the heart and blood vessels (e.g. heart failure, heart attack and stroke).

The main objective of the present study is to assess adherence to the IDC intervention and, consequently, its effectiveness on the prevention of the above mentioned diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-65 years
* Presence of any cardiovascular risk factors (Hypertension, Hypercholesterolemia, tobacco smoking, diabetes, obesity)

Exclusion Criteria:

* Currently diagnosed with any vardiovascular disease
* Currently involved in any other clinical trial
* Cognitive impairment that prevents from providing an informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk as calculated by means of the SCORE (Systematic Coronary Risk Evaluation) scale. Low-risk regions version. | upt to 12 months from the beginning

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline, 6 and 12 months from the beginning
  Spanish version of the EQ-5D-5L questionnaire by the EuroQol Group

OTHER OUTCOMES:
Chronic low-grade inflammation | Baseline, 6 and 12 months from the beginning
  High sensibility c-reactive protein